CLINICAL TRIAL: NCT04538651
Title: A Cross-sectional Study for Renal Function of Patients With Chronic Hepatitis B in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, Associate Professor, Sun Yat-sen University
Other Study IDs: XC3
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis B, Chronic
Keywords: renal function; chronic hepatitis B; antiviral treatment
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To acknowledge the prevalence of renal insufficiency and kidney-related diseases in patients with chronic hepatitis B in China through epidemiological surveys in outpatient clinics of about 150 hospitals across the country; 2. To analyze the related factors of renal insufficiency and kidney-related diseases in domestic patients with chronic hepatitis B from the aspects of demographic characteristics, family history, antiviral treatment, nephrotoxic drug use history, etc.

DETAILED DESCRIPTION:
At present, the mainstream antiviral treatment of CHB is still nucleotide analogues. The increase in the proportion of comorbidities in patients with chronic hepatitis B also increases the risk of nucleotide analogue contraindications. The antiviral treatment of CHB patients needs to fully assess the risk of adverse reactions . Taking into account the current impact of nucleotide analogs on renal function, the AASLD 2018 Chronic Hepatitis B Guidelines recommends that the dosage of nucleotide analogs should be adjusted according to renal function and creatinine clearance. A Hong Kong cohort study of patients with chronic hepatitis B showed that the 5-year chronic kidney disease (CKD) progression rate of patients receiving entecavir and tenofovir and not receiving treatment reached 40%. A similar study in the United States also showed that nucleotide analogs reduce the glomerular filtration rate (estimated glomerular filtration rate, eGFR). Studies on the indicators of early kidney injury found that the β2 microglobulin and retinol binding protein indicators changed significantly during the course of patients receiving adefovir dipivoxil, and the baseline β2 microglobulin and retinol binding protein indicators Affect the reduction of eGFR. Retrospective analysis using recent domestic urban medical insurance data also observed that the proportion of chronic kidney disease diagnoses in domestic CHB patients has shown a significant upward trend, which also suggests the necessity of assessing renal function in domestic CHB patients before using nucleotide analogs. Due to the lack of real-world renal function screening studies for CHB patients in China, there is a risk of severe underestimation of the proportion of CHB patients with renal insufficiency estimated based on medical insurance data. In the real world, the proportion of domestic CHB patients with renal insufficiency has not been fully clarified. Domestic clinical The treatment guidelines also did not specifically emphasize the necessity of renal function assessment before receiving nucleotide analog treatment.

Therefore, the purpose of this study is to understand the prevalence of renal insufficiency among people receiving hepatitis B antiviral treatment through a national epidemiological cross-sectional survey, using hospital outpatient clinics as the research site, and to analyze related factors to improve clinicians Awareness of renal insufficiency in patients with CHB and better guidance on the safe use of nucleotide analogs in patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B who are older than 18 years old and younger than 75 years old;
* Currently receiving nucleotide antiviral therapy;
* Patients are willing to undergo laboratory tests related to renal function: renal function items include glomeruli Filtration rate (eGFR), urea nitrogen (BUN), blood creatinine, uric acid, beta 2 microglobulin, alpha 1 microglobulin and urine protein, etc.;
* The patient is willing to undergo blood glucose testing;
* The patients are informed and agree to participate in this session the study.

Exclusion Criteria:

* Patients with decompensated liver cirrhosis;
* Patients with HIV infection and malignant tumors;
* Patients with severe mental illness or unable to cooperate;
* Female patients during lactation and pregnancy;
* Participation within three weeks or present Those who are participating in clinical research of other new drugs;
* Those who cannot understand or express informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to ensure the representativeness of the research subjects, this study will be carried out in the liver disease clinics of about 150 participating hospitals across the country. The source of the hospitals will take into account the region, city size and compliance. After each hospital project is launched, the epidemiological investigation will be completed within 1-3 months according to the sample size allocated by each hospital.
Sampling Method: Probability Sample
Enrollment: 11453 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate（eGFR） | within 3 months before study inclusion
  The amount of ultrafiltrate produced by the kidneys on both sides per unit time (per minute), called glomerular filtration rate, is an important indicator of renal function. Clinically, the glomerular filtration rate estimated in combination with the patient's gender, age, weight, and creatinine value is called the estimated glomerular filtration rate.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Xie, PhD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided